CLINICAL TRIAL: NCT04476160
Title: Effectiveness of Cinnamon on Insulin Resistance and Corporate Composition of Obese Schoolchildren
Brief Title: Effectiveness of Cinnamon on Insulin Resistance ( ECIRCCOS ) December 1, 2019
Acronym: ECIRCCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Collaborators: Hospital Infantil de Mexico Federico Gomez (Other)
Responsible Party: Principal Investigator, Jessie Nallelly Zurita Cruz, principal investigator, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-2018-785-108
Record Dates: First submitted 2019-11-12; First posted 2020-07-17 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2020-07

CONDITIONS: Obesity, Childhood; Insulin Resistance; Insulin Sensitivity
MeSH Terms: conditions — Pediatric Obesity; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cinnamon (Experimental): In this group, children will receive an intervention with 3000mg / day cinnamon along with diet and physical activity recommendations according to the WHO guidelines. They will be followed for 16 weeks. During this period, patients will be contacted weekly to corroborate the consumption of the capsules and interrogation of adverse effects such as dyspepsia, gastrointestinal disturbances and headache. They will be scheduled monthly for capsule counting and interrogation of adverse effects.
  Interventions: Dietary Supplement: Cinnamon
- Control (No Intervention): In this group, children will receive a placebo intervention along with diet and physical activity recommendations according to the WHO guidelines. They will be followed for 16 weeks. During this period, patients will be contacted weekly to corroborate the consumption of the capsules and interrogation of adverse effects such as dyspepsia, gastrointestinal disturbances and headache. They will be scheduled monthly for capsule counting and interrogation of adverse effects.

INTERVENTIONS:
Dietary Supplement: Cinnamon — children recipe 3 grams by day of cinnamon
  Arms: Cinnamon

SUMMARY:
Childhood obesity is one of the most serious public health problems of the 21st century. It is considered that if there are no changes in prevention and treatment strategies there will be an increase to 70 million obese children by 2025. Of the only pharmacological treatments accepted at this age to improve insulin resistance is metformin, but it can condition gastrointestinal, muscular and hepatic adverse events. Cinnamon is an alternative therapy, which due to its high concentrations of polyphenols, improves insulin resistance by decreasing the proinflammatory environment that occurs in this group of patients, and unlike metformin with less frequent adverse events. The effectiveness of cinnamon has been demonstrated by decreasing insulin resistance in the adult population.

DETAILED DESCRIPTION:
Controlled clinical trial, 100 children aged 10 to 15 years with obesity Body Mass Index (BMI> 2 SD) will be selected. Children and parents who agree to participate will be measured anthropometry (weight, height, BMI, body fat) and Tanner stage. Once the 100 children have been selected and registered, a determination will be made after 8 hours of fasting leptin, ghrelin, insulin, lipid profile, liver function tests, creatinine and cinnamic acid. Subsequently they will be randomly assigned to a group that receives the intervention with cinnamon 3000mg / day, or placebo; Both groups will receive diet and physical activity recommendations according to the World Health Organization (WHO) guidelines. They will be followed for 16 weeks. During this period, patients will be contacted weekly to confirm the consumption of the capsules and interrogation of adverse effects such as dyspepsia, gastrointestinal disturbances and headache. They will be scheduled monthly for capsule counting and interrogation of adverse effects. At the end of the 16-week follow-up, anthropometry, fasting after 8 hours of leptin, ghrelin, insulin lipid profile, liver function tests, creatinine and cinnamic acid will be performed.

Statistical analysis: Shapiro Wilk test will be applied to the variables with quantitative measurement scale to identify the type of distribution; in the case of parametric distribution, the data with averages and standard deviation will be presented, in case of presenting non-parametric distribution, medium and minimum and maximum values will be used. In the case of qualitative variables, they will be expressed with percentages and simple frequencies. Baseline characteristics will be compared between the two groups with t-Student or U-Mann Whitney according to the type of distribution of the variables. To evaluate the effect of the intervention, body fat deltas and biochemical measurements will be calculated by subtracting the final value (after 16 weeks of intervention) from the initial (baseline) value and statistical significance will be evaluated using comparisons between groups with paired t- or Wilcoxon. Covariance analysis control of confounding variables (ANCOVA) will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* obesity (BMI > 95 percentile )

Exclusion Criteria:

* treatment with insulin or Metformin
* genetic or endocrine obesity
* routine consumption of cinnamon

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
homeostatic model assessment (HOMA) index | 16 weeks
  resistence insulin is evaluated for fasting glucose and insulin
Appetite hormone (ghrelin [pg/ml]) | 16 weeks
  Change in fasting serum ghrelin from baseline to the end of intervention
Appetite hormone (leptin [ng/ml]) | 16 weeks
  Change in fasting serum leptin from baseline to the end of intervention

SECONDARY OUTCOMES:
Body mass index (BMI) | 16 weeks
  change in BMI from baseline to the end of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jessie Nallelly Zurita Cruz, Principal Investigator — Coordinación de Investigación en Salud, México
Locations (2):
- Mexico (2):
  - Unit of research in Medical Nutricion, Pediatric Hospital CMN "Siglo XXI" , Instituto Mexicano del Seguro Social, México, México City
  - Instituto Mexicano del Seguro Social, Mexico City